CLINICAL TRIAL: NCT01538407
Title: A Study of Strengthening Exercise on Quadriceps Force During Walking
Brief Title: Strengthening Exercise and Quadriceps Force During Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Principal Investigator, Marius Henriksen, Senior Researcher, PT. PhD, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 117.0
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Knee Osteoarthritis
Keywords: Strength training; Biomechanics; Quadriceps; Gait
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No intervention group
- Strength training group (Active Comparator): The knee extension strength training intervention period is 12 weeks with training sessions three times per week.
  Interventions: Other: Strength Training

INTERVENTIONS:
Other: Strength Training — The exercises will be performed in standard strength training equipment. Prior to each of the strengthening exercise sessions, a warm up phase is performed by 5-10 minutes of ergometer cycling at a moderate intensity. Muscle strengthening exercises will be performed according to the standard progressive resistance and overload principle. The exercise programme consists of three exercises performed with three sets of 10 repetitions at 60%-85% of patient's 10RM. Training load will be progressed by means of bi-weekly estimates of muscle strength to ensure a constant load of 60%-85% RM. Exercises are: 1. Leg extension, 2. Leg press, and 3. Forward lunges.
  Arms: Strength training group

SUMMARY:
This is a longitudinal, randomized, controlled interventional multi centric study on the effects of lower leg strengthening exercise on quadriceps force during walking in people with knee osteoarthritis. At each study centre twenty subjects will be included, for a total of 40 participants. Subjects will be randomized equally (1:1) into 1 active arm and 1 control arm.

The objective of the study is to evaluate the effect of twelve weeks of quadriceps strengthening on the mechanical output of the quadriceps during locomotion. A secondary purpose is to explore the relationship between quadriceps strengthening and compressive knee loadings. The hypothesis is that quadriceps strength training will not change quadriceps force, power, and work in locomotion in people with knee osteoarthritis.

Primary outcome is quadriceps force during walking, secondary outputs are quadriceps power and work and knee compressive loads during walking. Explorative measures are isometric and concentric isokinetic leg muscle strength, radiographic score of the knee (Kellgren and Lawrence), a one-leg rise from chair test (maximum number of reps) and a lateral step-up test (maximum number of reps).

ELIGIBILITY:
Inclusion Criteria:

A medical doctor will perform the screening of potential participants. Subjects must meet the following inclusion criteria to be eligible for study entry:

* Knee OA diagnosed according to the American College of Rheumatology criteria (26), with clinical symptoms and radiographically verified tibio-femoral osteoarthritis in one or both knees.
* Aged between 40 and 65 yrs.
* Untrained (i.e. less than 2 hours of exercise per week)
* Subject must not be using assistive walking device
* Willing and able to complete study visits and procedures
* Willing to hold activity and exercise level generally consistent during the study except that encompassed in the study.
* In general good health, in the opinion of the investigator, based on medical history and physical examination and, if necessary, laboratory values. Laboratory tests are prescribed by the medical doctor at the screening visit.
* A body mass index (BMI) of 19<BMI≤32kg/m2
* Speaks, reads and writes Danish and/or English language

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria will be ineligible for study entry:

* Subjects depending on walking device
* Pregnant or breastfeeding
* Radiographic evidence of Patello-femoral knee OA only (and no tibio-femoral OA).
* History of symptoms of autoimmune disorders (e.g., inflammatory bowel disease, multiple sclerosis, lupus, rheumatoid arthritis)
* Planned surgical procedure during the duration of the study
* History or diagnosis of musculoskeletal injuries or pathologies, including but not limited to:

  * Anterior cruciate ligament injuries
  * Meniscal injuries related to trauma (degenerative changes allowed)
  * Patellofemoral Pain Syndrome
  * Low back pain
* History, diagnosis, or signs and symptoms of clinically significant cardiovascular disease, including but not limited to:

  * Ischemic heart disease
  * Arthrosclerosis
  * Peripheral artery disease
* History, diagnosis, or signs and symptoms of diabetes
* History, diagnosis, or signs and symptoms of neurological disorders including but not limited to

  * Stroke
  * Parkinson's disease
  * Multiple sclerosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in peak quadriceps force during walking at 12 weeks | Baseline and at 12 weeks
  Estimates of the quadriceps muscle forces during locomotion are calculated using a biomechanical model based on data from gait analysis

SECONDARY OUTCOMES:
Change from baseline in quadriceps power and work during walking at 12 weeks | Baseline and after 12 weeks
  Estimated from gait analysis
Change from baseline in knee compressive force during walking at 12 weeks | Baseline and after 12 weeks
  Estimated from biomechanical modelling of data from gait analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Devita, MSc, PhD, Principal Investigator — The College of Health and Human Performance, Department of Exercise and Sport Science, Minges Coliseum Greenville, U.S.A.; Marius Henriksen, PhD, Study Director — The Parker Institute, Frederiksberg University Hospital
Locations (2):
- The College of Health and Human Performance, Department of Exercise and Sport Science, Minges Coliseum, Greenville, North Carolina, United States
- The Parker Institute, Frederiksberg University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] DeVita P, Aaboe J, Bartholdy C, Leonardis JM, Bliddal H, Henriksen M. Quadriceps-strengthening exercise and quadriceps and knee biomechanics during walking in knee osteoarthritis: A two-centre randomized controlled trial. Clin Biomech (Bristol). 2018 Nov;59:199-206. doi: 10.1016/j.clinbiomech.2018.09.016. Epub 2018 Sep 15. PMID 30273922